CLINICAL TRIAL: NCT03914469
Title: MOTIVATE: Moving to Improve Chronic Back Pain and Depression in Older Adults
Brief Title: MOTIVATE: Moving to Improve Outcomes for Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to poor recruitment.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Una Makris, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU 2018-0084
Record Dates: First submitted 2019-04-01; First posted 2019-04-16 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Back Pain Lower Back Chronic

STUDY DESIGN:
Intervention Model Description: Investigators will assess the feasibility of a tele-delivered behavioral change intervention among older adults (aged 50 and older) with cLBP and depression. Fifty participants will be randomly assigned to one of two groups, behavioral intervention arm (n=25) versus the waitlist control arm (n=25).
Who Masked: Outcomes Assessor
Masking Description: The research staff conducting outcomes assessments will be blinded to whether the subject is in active or waitlist group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control Group (No Intervention): The waitlist control group will continue with management of chronic back pain and depression per usual care. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, mid-point, final assessments) conducted by a blinded research assistant. Subjects randomized to the waitlist control group will be offered the same intervention once the active intervention group has completed the active sessions and assessments.
- Behavioral Intervention Group (Experimental): For participants assigned to the intervention arm, trained health coaches will deliver the intervention via telephone. All participants, regardless of what group they have been assigned to will undergo several outcome assessments (pre-screening, baseline, mid-point, final assessments) conducted by a blinded research assistant.
  Interventions: Behavioral: Behavioral Intervention Group

INTERVENTIONS:
Behavioral: Behavioral Intervention Group — The active intervention will include eight tele-delivered health coach sessions, three tele-based outcome assessments, and up to two semi-structured interviews at 6 months post-intervention. Each tele-based outcome assessment is roughly 45-60 minutes and will be conducted by a member of the research team. Each intervention session will be delivered by a trained health coach over a period of 10-20 weeks (up to 5 months total, accounting for additional time between sessions if needed).
  Arms: Behavioral Intervention Group

SUMMARY:
The overarching goal of this study is to evaluate a tele-based behavioral change intervention for older adults (aged 50 years and older) with chronic low back pain (cLBP) and comorbid depression, and to ultimately assess its effect on cLBP-related disability and depressive symptoms.

Investigators will conduct a pilot randomized control trial to assess feasibility for older adults with chronic low back pain and depression to receive a behavioral change tele-based intervention delivered by a health coach trained in motivational interviewing. All participants, regardless of intervention arm assigned, will undergo outcomes assessments (baseline, mid-point, final assessments) conducted by a blinded research assistant.

DETAILED DESCRIPTION:
Investigators will assess the feasibility of a tele-delivered behavioral change intervention among older adults (aged 50 and older) with chronic low back pain and depression. Fifty participants will be randomly assigned to one of two groups, behavioral intervention arm (n=25) versus the waitlist control arm (n=25). The active intervention will include eight tele-delivered health coach sessions, three tele-based outcome assessments, and up to two semi-structured interviews within 6 months of completion, post-intervention. Each tele-based outcome assessment is roughly 45-60 minutes and will be conducted by a member of the research team. Each intervention session will be delivered by a trained health coach over a period of 10-20 weeks (up to 5 months total, accounting for additional time between sessions if needed).

The first session will introduce the participant to the health coach and the program, establish rapport, and measure baseline physical activity. The following six sessions address behavioral determinants, followed by a final session designed to be a booster session to the overall program.

An Omron pedometer will be provided to each participant for the assessment of physical activity. The Omron pedometer will be set up by a member of the research team (e.g., stride length, setting date/time) and will be mailed to the participant's home address between sessions one and two. Each participant will receive a courtesy phone call when the pedometer is mailed and will be asked to call the research coordinator when it arrives. The research team will provide technical assistance and instructions to the participant regarding use. The pedometer is intended to be worn on the waist band, daily, with the exception of times when the participant may shower or bathe. The research team will verbally instruct the participant on how to press the mode and memory buttons in order to provide weekly step counts for tracking physical activity. The participants will be prompted by the health coach or research staff to report step counts during subsequent weekly tele-based coaching sessions.

Since the investigators are interested in better understanding feasibility of the intervention as compared to the waitlist control, and how behaviors are sustained over time, the study involves follow-up to 6 months. Investigators will use these follow-up data to better understand differential attrition as well as preliminary formative implementation evaluation. Using purposive sampling, investigators will conduct ~ 10 in-depth semi-structured interviews. Each interview will occur ~six months post-intervention and will include key stakeholders from the following groups: study participants from each arm of the pilot study, the health coach, primary care and mental health providers.

The research staff will select participants identified as higher risk for drop-out, less engaged, or were particularly successful at achieving behavioral change. The purpose of the final interviews is to learn about the barriers and facilitators to successful intervention delivery and participant retention from the perspectives of the enrolled patients, health coach, and providers. Interview topics will borrow from components of the well-established framework, Promoting Action on Research Implementation in Health Services (PARiHS). Semi-structured interview strategy is informed by two Promoting Action on Research Implementation in Health Services (PARiHS) dimensions: context-how the microsystem (UTSW) impacts behavioral change uptake, for example, potential facilitators to intervention implementation; facilitation-identifying specific ways to augment the likelihood of implementation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 and older
* English- speaking
* Working telephone
* Capable of participating in home-based activity
* Chronic low back pain with intensity of 4 or higher on 10 point scale
* Self-reported low back pain (+/-radiation) in the past 3 months that interferes with daily activities on most days
* Depression, PHQ-9>10 stable (per chart review, no psychotic or suicidal ideation; confirmed over telephone)

Exclusion Criteria:

* Aged 49 or less
* No telephone
* Not English speaking
* Unwilling to be randomized to either study arm
* Self-reported, uncorrected hearing or visual disturbance precluding ability to participate in telephone sessions or read pedometer screen
* Cognitive impairment, assessed by Memory Impairment Screen
* Lumbar surgery within the last year
* Self-reported dependence on wheelchair, bed-bound, or severe balance impairment (unable to participate in physical activity intervention)
* Illness requiring hospitalization within the last 3 months (e.g., fall, gout attacks, stroke, heart attack, heart failure, or surgery for blocked arteries)
* Suicidal ideation or prior psychotic episodes requiring hospitalization within the last year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Una Makris, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health & Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Started | 6 | 6
Completed | 5 | 2
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control Group | Behavioral Intervention Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66.8 [53 to 81] | 59.0 [51 to 67] | 62.9 [51 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rates
Description: Of patients pre-screened, the total number enrolled into the study
Time Frame: Through study completion, up to 6 months
Population: We pre-screened 371 participants and enrolled 12 (6 in each study arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 185 | 186
Participants | 6 | 6

2. Primary Outcome: Rate of Intervention Completion
Description: Of patients randomized into the intervention arm, the total number retained for follow-up
Time Frame: Through study completion, up to 6 months
Population: Of the 6 waitlist control arm participants, 5 completed assessments Of the 6 active behavioral intervention arm participants, 2 completed the program and assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 6 | 6
Participants | 5 | 2

3. Secondary Outcome: Pain Scale
Description: Pain intensity on 0-10 scale where higher values are worse pain. The data reported is the averaged data for the end assessments.
Time Frame: at approximately 4 months
Population: The study personnel entering data for the pain scale clicked some incorrect options that caused calculation errors preventing the assessment of the collected data or caused loss of data for 1 participant in the control group and hence it is not used in the analysis/reporting of this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 4 | 2
score on a scale | 4.8 (3.44) | 5.7 (0.67)

4. Secondary Outcome: Roland Morris Disability Questionnaire (RMDQ)
Description: Disability related to back pain. Scale ranges from 0-24 with larger numbers indicating worse disability related to chronic back pain. The data reported is the averaged data for the end assessments.
Time Frame: at approximately 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 5 | 2
score on a scale | 14.6 (5.43) | 10 (1)

5. Secondary Outcome: Depression
Description: Depression: Patient Health Questionnaire (PHQ-9) scored between 0-27 with higher numbers indicated worse depression. The data reported is the averaged data for the end assessments.
Time Frame: at approximately 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 5 | 2
score on a scale | 11.2 (6.62) | 18.5 (0.5)

6. Secondary Outcome: Step Counts
Description: Physical activity: step counts measured using Omron pedometer. Participants will wear the pedometer clipped to their right lateral waistband for 24 hours per day for 7 consecutive days (except during shower or water activities) to obtain 5 complete days of physical activity data. The data reported is the averaged data for session 8 of the intervention for each participant, among those who stayed in the study for all sessions.
Time Frame: at approximately 3 months
Population: Per protocol, only participants in the active arm received pedometers to report step counts. Therefore, step count data is only available for participants in the Behavioral Intervention Group that was analyzed and reported for this outcome measure.
Measure: Mean (Standard Deviation); unit: step counts
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
Number analyzed (Participants) | 0 | 3
step counts |  | 30102.33 (2138.03)

ADVERSE EVENTS:
Time Frame: Adverse event reporting from enrollment to end of study (typically 6 months)
Arm/Group | Waitlist Control Group | Behavioral Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Due to poor recruitment and early termination of this study, the collected data for the limited enrolled participants were not considered valid for any useful assessment for outcomes#3-6. Hence, these outcomes were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03914469/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03914469/ICF_001.pdf